CLINICAL TRIAL: NCT05550025
Title: A Single-center, Prospective, Single-arm Phase II Clinical Study on the Efficacy and Safety of TACE Combined With Camrelizumab and Apatinib in the Treatment of Advanced Liver Cancer
Brief Title: TACE Combined With Camrelizumab and Apatinib in the Treatment of Advanced Liver Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, xulinfeng, Director of Interventional Department, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-KY-195
Record Dates: First submitted 2022-07-25; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE combined with Apatinib and Camrelizumab (Experimental): TACE（transcatheter arterial chemoembolization） combined with Apatinib and Camrelizumab
  Interventions: Drug: camrelizumab& apatinib

INTERVENTIONS:
Drug: camrelizumab& apatinib — TACE（transcatheter arterial chemoembolization） combined with Apatinib and Camrelizumab Camrelizumab 200mg every 3 weeks. Taking Apatinib-Mesylate Tablets (250 mg/tablet) orally after meals, once a day, for continuous medication.
  The cumulative maximum drug use period is up to 1 years. The patient is concurrent on medication until the treatment discontinuation criteria specified in the protocol appear.

SUMMARY:
This study was designed to evaluate the effectiveness and safety of TACE（transcatheter arterial chemoembolization） combined with Apatinib and Camrelizumab for Hepatocellular Carcinoma.

The primary outcome measure is to evaluate the objective response rate (ORR) of the therapy for Hepatocellular Carcinoma.

The secondary Outcome measures include the duration of response (DOR), disease control rate (DCR), progression-free survival rate (PFSR) [ Time Frame: 6- and 12-month], overall survival rate (OSR) [ Time Frame: 6- and 12-month], the median progression-free survival time (mPFS) and median overall survival time (mOS) of the therapy for Hepatocellular Carcinoma.

Moreover, this study aims to assess the safety and tolerability of the Therapy for Hepatocellular Carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma is a common high-grade malignant tumor in my country, with limited treatment options and poor prognosis. Transcatheter arterial chemoembolization (TACE) is currently recognized as an effective method for the treatment of unresectable hepatocellular carcinoma. Intra-arterial administration and embolization are the two major features of TACE treatment techniques. However, conventional TACE (conventional TACE, CTACE) mainly focuses on the efficacy of embolization, and the effect of chemotherapy is not ideal. The emergence of drug-eluting beads (DEB) enhances the effect of chemotherapy in TACE, which is of great significance to improve the overall efficacy of TACE in hepatocellular carcinoma. However, the long-term efficacy of TACE in the treatment of liver cancer is not very satisfactory. Changes in the tumor microenvironment after TACE can induce abnormally elevated expression of tumor progression-related factors, which makes liver cancer cells prone to local recurrence and distant metastasis, which seriously affects the prognosis of liver cancer patients. Clinical studies have shown that the complete tumor necrosis rate of TACE treatment of liver cancer is only 10-20%, and the median survival time of patients is only 16-20 months. Therefore, the poor long-term efficacy of TACE is an urgent bottleneck for its application in the clinical treatment of liver cancer.

With the deepening of tumor immune theory research, based on overcoming the immune escape of swelling and pain, the therapy that produces a specific and efficient immune response to swelling and pain has gradually become a hot spot in tumor research, and great progress has been made. Tumor immunotherapy has the advantages of high specificity, remarkable curative effect, and slight damage to normal organisms.The 2018 Nobel Prize in Physiology or Medicine was awarded to American scientist James R Alison and Japanese scientist Tasuku Honjo for their pioneering contributions to tumor immunotherapy. With the in-depth study of the theory of swelling and pain immunology and the continuous progress of treatment technology, it is expected to achieve a new breakthrough in the radical cure of swelling and pain, and has gradually become the mainstream method of tumor treatment.

Programmed death 1 (PD-1)/programmed death-ligand 1 (PD-L1) signaling pathway is currently the most mature and fastest-growing tumor immunotherapy molecule target. PD-1 plays a role in the effector phase of the immune response and is expressed on activated T cells, B cells and myeloid cells. PD-1 has two ligands, namely PD-L1 and PD-L2. Both PD-L1/L2 are expressed in antigen-presenting cells, and PD-L1 is also expressed in various tumor tissues. The combination of PD-1 and PD-L1 mediates the co-inhibitory signal of T cell activation, inhibits the killing function of T cells, and negatively regulates the human immune response. Therefore, immunomodulation targeting PD-1/PD-L1 is of great significance for anti-tumor therapy.

Camrelizumab is a humanized PD-1 monoclonal antibody independently developed by Jiangsu Hengrui Medicine. It has completed a phase clinical study for the treatment of solid pain. The results show that camrelizumab has the potential to treat advanced solid pain. Good safety and tolerability. Objective response rate of camrelizumab in patients with previously treated advanced hepatocellular carcinoma. A multi-center clinical trial of patients who received at least TACE. Combination with camrelizumab and apatinib in the treatment of advanced liver tumors. A single-center, pre-fragile, single-arm, phase I clinical study Among patients receiving first-line systemic therapy, the 6-month overall survival rate was 74.4% (95%CI.68.0-79.7), with anti-swelling and pain activity, and the safety was controllable, so camrelizumab was approved for liver cancer indications on March 6, 2020 , for patients with advanced hepatocellular carcinoma who have previously received sorafenib and/or oxaliplatin-containing 14.7%(95%CI 10.3-20.2), systemic chemotherapy.

Apatinib is a new-generation small-molecule vascular endothelial growth factor receptor-2 (VEGFR-2) tyrosine kinase inhibitor, and the world's first small-molecule anti-angiogenic target proven safe and effective in the treatment of advanced gastric cancer Xiang drug, independently developed by Jiangsu Hengrui Medicine, its main mechanism of action is to highly selectively inhibit the signal transduction of VEGFR-2 combined with the micro-activity of succinic acid, yang-blocking vascular endothelial growth factor (VEGF), thereby effectively inhibiting the Swelling angiogenesis. In 2020, the "randomized, bilingual, placebo-controlled phase W AHELP study of second-line apalachone in the treatment of late Ming hepatocellular brain (CHCC)" jointly conducted by 31 tumor centers across the country" was accepted by the ASCO General Assembly and selected as an oral presentation. The results of the study showed that, compared with placebo, apatinib significantly prolonged median OS in previously treated Chinese patients with advanced HCC (8.7 months vs 6.8 months). In addition, the median progression-free survival (PFS) in the apatinib group was 4.5 months, compared with 19 months in the placebo group. at the same time, the objective response rate (ORR) of the apatinib group was 10.7%, which was significantly higher than that of the control group of 1.5%. In terms of safety, treatment-related adverse events were similar to those already approved for the treatment of late-stage gastric cancer, no new adverse events were observed, and patients were well tolerated. Although apatinib has been submitted to the CFDA for second-line indications for hepatocellular carcinoma, it has not yet been officially approved, so it has not been written in the instructions, that is, it is an off-label drug.

A phased study of apalacone combined with transarterial chemoembolization (TACE) in the treatment of advanced liver cancer was published in the journal Cancer Biology & Therapy. Preliminary conclusions showed that apazatinib combined with TACE treatment significantly improved ORR at 9 and 12 months, and the median PFS was also significantly better than the control group (12.5 months vs. .6.0 months). Another single-center retrospective study also confirmed that, the PFS and OS of apalacone combined with TACE in the treatment of advanced liver tumors were significantly better than those of the control group. It can be seen that combined with apatinib treatment on the basis of TACE, hopefully better Inhibit the growth of swelling disease to prolong the disease-free survival period and improve the survival rate of patients. In 2018, a retrospective study was published at the World Congress on Pain and Pain Intervention (WCIO), suggesting the survival benefit of apalacone combined with TACE in the treatment of patients with HCC and portal vein tumor thrombus (PVTT). Apatinib combined with camrelizumab in the treatment of advanced liver cancer, gastric cancer and esophagogastric junction cancer! The phase clinical study also showed the synergistic effect of immunotherapy and anti-angiogenic therapy, of which 16 cases of liver cancer can be evaluated for efficacy, ORR and DCR were 50% and 93.8%, respectively. The results of the study were presented at the ASCO. Annual meeting. Apatinib in combination with camrelizumab for advanced liver cancer due to encouraging findings Phase clinical research is also actively carried out, and all subjects have now been enrolled. At the same time, a single-center study on the efficacy and safety of apatinib combined with camrelizumab versus sorafenib in the first-line treatment of advanced hepatocyte TACE combined with camrelizumab and apatinib in the treatment of advanced liver cancer , Prospective, single-arm, Phase II clinical trials of cancer cells in Sichuan have also been launched simultaneously in China, the United States, and Europe. This randomized, controlled, open-label, international multi-center study is the first exploration of the combination of PD-1 monoclonal antibody and anti-vascular targeting in my country in the field of liver cancer in the world. We look forward to the announcement of the follow-up research results.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, ≤ 70 years old, both men and women;
2. Clinical or pathologically confirmed BCLC C-stage hepatocellular carcinoma, no further first-line treatment;
3. At least one intrahepatic evaluable tumor existed, intrahepatic tumor is the primary tumor burden;
4. Child-Pugh score small or equal to 7 points (Child-Pugh A-B);
5. The liver tumor burden does not exceed 50% of the total liver volume;
6. Patient can swallow tablet normally;
7. ECOG score: 0 to 1 (according to the ECOG score classification);
8. The expected survival is longer than 12 weeks;

Exclusion Criteria:

1. The patient has any active auto-immune disease or a history of auto-immune disease (such as the following, but not limited to: auto-immune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, thyroid hyperfunction; patients with vitiligo. For patient with history of asthma, complete remission of asthma in childhood without any intervention after adulthood can be included, while those asthma patients who require bronchodilators for medical intervention cannot be included.);
2. The patient is using immunosuppressive agents or systemic hormonal therapy for immunosuppression purposes (dose > 10 mg/day of prednisone or other therapeutic hormones) and continues to be used within 2 weeks prior to enrollment;
3. Severe allergic reactions to other monoclonal antibodies;
4. Known for a history of central nervous system metastasis or hepatic encephalopathy;
5. Having a history of organ transplantation;
6. Patients with clinically symptomatic ascites who require puncture, drainage, or ascites drainage within 3 months, except for those who have a small amount of ascites but no clinical symptoms;
7. Suffering from hypertension, and cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥ 140mmHg or diastolic blood pressure ≥90 mmHg);
8. Suffering heart diseases with clinical symptoms or those not well controlled, such as: (1) heart failure in NYHA class 2 or higher; (2) unstable angina; (3) myocardial infarction occurred within 1 year; (4) clinically symptomatic supraventricular or ventricular arrhythmia requiring treatment or intervention; (5) Tc > 450ms (male); QTc > 470ms (female);
9. Coagulation dysfunction (INR>2.0, PT>16s), bleeding tendency or receiving thrombolysis or anticoagulant therapy, allowing prophylactic use of low-dose aspirin or low molecular heparin;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2023-11-11 (Estimated); Study Completion 2024-02-11 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST 1.1 and mRECIST | From date of first dose of study drug until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to approximately 3 years)
  ORR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) at the time of data cutoff as assessed by RECIST 1.1 and mRECIST

SECONDARY OUTCOMES:
The median overall survival time (mOS) | From the start date of the Treatment Phase until date of death from any cause (up to approximately 3 years)
  OS is measured from the start date of the Treatment Phase (date of first study dose) until date of death from any cause. Participants who are lost to follow-up and the participants who are alive at the date of data cutoff will be censored at the date the participant was last known alive or the cut-off date, whichever comes earlier.

CONTACTS AND LOCATIONS:
Overall Officials: xu Linfeng, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No